CLINICAL TRIAL: NCT00719797
Title: A PHASE III RANDOMIZED TRIAL OF FOLFOXIRI + BEVACIZUMAB VERSUS FOLFIRI + BEVACIZUMAB AS FIRST- LINE TREATMENT FOR METASTATIC COLORECTAL CANCER
Brief Title: Combination Chemotherapy and Bevacizumab as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Acronym: TRIBE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000598582; GONO-TRIBE; ASL608LIOM04; EUDRACT:2008-001537-10
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV rectal cancer; stage IV colon cancer; stage III rectal cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (FOLFOXIRI) (Experimental): Patients receive irinotecan hydrochloride IV over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (FOLFIRI) (Experimental): Patients receive irinotecan hydrochloride IV over 1 hour, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: bevacizumab — Given IV
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV
  Arms: Arm I (FOLFOXIRI)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This randomized phase III trial is comparing two combination chemotherapy regimens given together with bevacizumab to see how well they work as first-line therapy in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of bevacizumab in combination with oxaliplatin, irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFOXIRI) versus bevacizumab in combination with irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFIRI) in patients with unresectable, metastatic colorectal cancer.

Secondary

* To evaluate the safety profile, including long-term adverse events of these regimens in these patients.
* To compare the overall response rate, duration of response, and secondary R0 surgery rates of metastases and overall survival between treatment arms.
* To evaluate potential surrogate markers predictive of bevacizumab activity.

OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status (0 vs 1-2), prior adjuvant chemotherapy (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (FOLFOXIRI): Patients receive irinotecan hydrochloride IV over 1 hour, oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.
* Arm II (FOLFIRI): Patients receive irinotecan hydrochloride IV over 1 hour, leucovorin calcium IV over 2 hours, and bevacizumab IV on day 1. Patients also receive fluorouracil IV continuously over 48 hours beginning on day 1.

In both arms, treatment repeats every 2 weeks for up to 12 courses. Treatment with bevacizumab, fluorouracil, and leucovorin calcium continues in the absence of disease progression or unacceptable toxicity.

Patients undergo serum extraction and blood sample collection periodically for genotyping studies. Patients also undergo collection of tumoral sections from paraffin embedded primary and/or metastatic lesions periodically for immunohistochemical analyses.

After completion of study treatment, patients are followed every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Unresectable metastatic disease
* Measurable disease, defined as ≥ 1 measurable lesion according to RECIST criteria
* No prior chemotherapy for metastatic disease
* No untreated brain metastases, spinal cord compression, or primary brain tumors
* No history or evidence of CNS disease by physical examination unless adequately treated (e.g., uncontrolled seizure despite standard medical therapy or history of stroke)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-2 (≤ 70 years of age) OR ECOG PS 0 (71-75 years of age)
* Life expectancy ≥ 12 weeks
* Neutrophils ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin > 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN if f liver metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN if liver metastases present)
* Creatinine clearance > 50 mL/min OR serum creatinine ≤ 1.5 times ULN
* Proteinuria < 2+ by dipstick OR urine protein ≤ 1 g by 24-hr urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled hypertension
* Clinically significant (i.e., active) cardiovascular disease, including any of the following:

  * Cerebrovascular accidents within the past 6 months
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
* Known allergy to Chinese hamster ovary cell proteins or any of the components of the study medications
* Other co-existing malignancy or malignancy diagnosed within the past 5 years, except for basal cell or squamous cell carcinoma, or carcinoma in situ of the cervix
* Symptomatic peripheral neuropathy ≥ grade 1 according to the NCI Common Toxicity Criteria
* Lack of physical integrity of the upper gastrointestinal tract
* Malabsorption syndrome
* Inability to take oral medication
* Significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* More than 10 days since prior and no concurrent ongoing treatment with anticoagulants for therapeutic purposes
* More than 28 days since prior and no concurrent major surgical procedure
* More than 28 days since prior open biopsy
* More than 30 days since prior investigational agents
* No concurrent chronic daily high-dose acetylsalicylic acid (> 325 mg/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival | up to 54 months
  To compare the progression free survival of bevacizumab in combination with oxaliplatin, irinotecan and infusional 5FU/LV ("GONO" FOLFOXIRI regimen) to bevacizumab in combination with irinotecan and infusional 5FU/LV (FOLFIRI regimen)

SECONDARY OUTCOMES:
Overall response rate | up to 54 months
Duration of response | up to 54 months
Secondary R0 surgery rates of metastases | up to 54 months
Overall survival | up to 54 months
Surrogate markers predictive of bevacizumab activity | up to 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Presidio Ospedaliero di Livorno
Locations (44):
- Italy (44):
  - Ospedale Civile Ss. Antonio E Biagio Di Alessandria - Alessandria (Al) Oncologia Medica, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona - Ancona (An) Oncologia Medica, Ancona
  - P.O. Zona Aretina - Ospedale S. Donato Di Arezzo - Arezzo (Ar) Oncologia Medica, Arezzo
  - Irccs Centro Di Riferimento Oncologico (Cro) - Aviano (Pn) Oncologia Medica, Aviano
  - Ospedale S. Orsola F.B.F. - Brescia - Brescia (Bs) Oncologia Medica, Brescia
  - Istituto Ospedaliero Fondazione Poliambulanza Di Brescia - Brescia (Bs) Oncologia Medica, Brescia
  - Stabilimento "Perrino" - Brindisi - Brindisi (Br) Oncologia Medica, Brindisi
  - Azienda Ospedaliera S. Elia - Caltanissetta (Cl) Oncologia Medica, Caltanissetta
  - Ausl 1 Di Massa E Carrara - Carrara (Ms) Oncologia Medica, Carrara
  - Ospedale Cecina - Cecina (Li) Oncologia Medica, Cecina
  - Istituti Ospitalieri - Cremona - Cremona (Cr) Oncologia Medica, Cremona
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo - Cuneo (Cn) Oncoematologia, Cuneo
  - Ausl 11 Di Empoli (Fi) - Empoli (Fi) Oncologia Medica, Empoli
  - U.S.L.N.6 -Ospedale Civile 'E.Profili'-F - Fabriano (An) Oncologia Medica, Fabriano
  - Ausl 10 Di Firenze - Firenze (Fi) Oncologia Medica, Florence
  - Irccs Istituto Nazionale Per La Ricerca Sul Cancro (Ist) - Genova (Ge) Oncologia Medica, Genova
  - Ausl Le Di Lecce - Lecce (Le) Oncologia Medica, Lecce
  - Aulss 21 Di Legnago (Vr) - Legnago (Vr) Oncologia Medica, Legnano
  - Ausl 12 Di Viareggio (Lu) - Lido Di Camaiore (Lu) Oncologia Medica, Lido di Camaiore
  - Ospedale Livorno - Livorno (Li), Oncologia Medica, Livorno
  - Presidio Ospedaliero Piana Di Lucca - Lucca (Lu) Oncologia Medica, Lucca
  - Irccs Fondazione Centro S. Raffaele Del Monte Tabor - Milano (Mi) Oncologia Medica, Milan
  - Ospedale Ca' Granda-Niguarda - Milano - Milano (Mi) Oncologia Medica, Milan
  - S.Gerardo - Monza - Monza (Mi) Oncologia Medica, Monza
  - A.O. Universitaria Federico Ii Di Napoli Oncologia Medica, Napoli
  - A.O. Universitaria Maggiore Della Carita' Di Novara Oncologia Medica, Novara
  - A.O. Universitaria Di Parma Oncologia Medica, Parma
  - Asl 1 Di Citta' Di Castello (Pg) - Citta' Di Castello (Pg) Oncologia Medica, Perugia
  - A.O. Di Perugia - Ospedale S. Maria Della Misericordia (Ex Silvestrini) - Perugia (Pg) Oncologia Medica, Perugia
  - Azienda Ospedaliera San Salvatore - Pesaro (Pu) Oncologia Medica, Pesaro
  - Ospedale Della Valdinievole - Pescia (Pt) Oncologia Medica, Pescia
  - Ospedale Piombino - Piombino (Li) Oncologia Medica, Piombino
  - A.O. Universitaria Pisana Oncologia Medica, Pisa
  - Ausl 5 Di Pisa - Pisa (Pi) Oncologia Medica, Pisa
  - Alfredo Falcone A.O. Universitaria Pisana - Pisa (Pi) Oncologia Medica, Pisa
  - Ausl 3 Di Pistoia - Pistoia (Pt) Oncologia Medica, Pistoia
  - Ausl 4 Di Prato - Prato (Po) Oncologia Medica, Prato
  - Ospedale Di S. Maria Nuova - Reggio Nell'Emilia (Re) Oncologia Medica, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico Di Roma Oncologia Medica, Rome
  - Policlinico Umberto I Di Roma Oncologia Medica, Rome
  - Policlinico Universitario Gemelli Di Roma Oncologia Medica, Rome
  - A.O. Universitaria Senese Oncologia Medica, Siena
  - Ospedale Civile - Sondrio - Sondrio (So) Oncologia Medica, Sondrio
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino Oncologia Medica, Torino

REFERENCES:
- [Derived] Rossini D, Germani MM, Lonardi S, Pietrantonio F, Dell'Aquila E, Borelli B, Allegrini G, Maddalena G, Randon G, Marmorino F, Zaniboni A, Buonadonna A, Boccaccino A, Conca V, Antoniotti C, Passardi A, Masi G, Cremolini C. Treatments after second progression in metastatic colorectal cancer: A pooled analysis of the TRIBE and TRIBE2 studies. Eur J Cancer. 2022 Jul;170:64-72. doi: 10.1016/j.ejca.2022.04.019. Epub 2022 May 17. PMID 35594613
- [Derived] Antoniotti C, Germani MM, Rossini D, Lonardi S, Pietrantonio F, Santini D, Marmorino F, Allegrini G, Daniel F, Raimondi A, Borelli B, Zaniboni A, Conca V, Abraham J, Spetzler D, Maiello E, Boccaccino A, Passardi A, Giordano M, Tamburini E, Korn MW, Masi G, Cremolini C. FOLFOXIRI and bevacizumab in patients with early-onset metastatic colorectal cancer. A pooled analysis of TRIBE and TRIBE2 studies. Eur J Cancer. 2022 May;167:23-31. doi: 10.1016/j.ejca.2022.02.031. Epub 2022 Mar 30. PMID 35366570
- [Derived] Cremolini C, Antoniotti C, Stein A, Bendell J, Gruenberger T, Rossini D, Masi G, Ongaro E, Hurwitz H, Falcone A, Schmoll HJ, Di Maio M. Individual Patient Data Meta-Analysis of FOLFOXIRI Plus Bevacizumab Versus Doublets Plus Bevacizumab as Initial Therapy of Unresectable Metastatic Colorectal Cancer. J Clin Oncol. 2020 Aug 20:JCO2001225. doi: 10.1200/JCO.20.01225. Online ahead of print. PMID 32816630
- [Derived] Tokunaga R, Cao S, Naseem M, Lo JH, Battaglin F, Puccini A, Berger MD, Soni S, Millstein J, Zhang W, Stintzing S, Loupakis F, Cremolini C, Heinemann V, Falcone A, Lenz HJ. Prognostic Effect of Adenosine-related Genetic Variants in Metastatic Colorectal Cancer Treated With Bevacizumab-based Chemotherapy. Clin Colorectal Cancer. 2019 Mar;18(1):e8-e19. doi: 10.1016/j.clcc.2018.09.003. Epub 2018 Sep 13. PMID 30293873
- [Derived] Cremolini C, Antoniotti C, Lonardi S, Bergamo F, Cortesi E, Tomasello G, Moretto R, Ronzoni M, Racca P, Loupakis F, Zaniboni A, Tonini G, Buonadonna A, Marmorino F, Allegrini G, Granetto C, Masi G, Zagonel V, Sensi E, Fontanini G, Boni L, Falcone A. Primary tumor sidedness and benefit from FOLFOXIRI plus bevacizumab as initial therapy for metastatic colorectal cancer. Retrospective analysis of the TRIBE trial by GONO. Ann Oncol. 2018 Jul;29(7):1528-1534. doi: 10.1093/annonc/mdy140. Epub 2018 Apr 20. PMID 29873679
- [Derived] Cremolini C, Del Re M, Antoniotti C, Lonardi S, Bergamo F, Loupakis F, Borelli B, Marmorino F, Citi V, Cortesi E, Moretto R, Ronzoni M, Tomasello G, Zaniboni A, Racca P, Buonadonna A, Allegrini G, Ricci V, Di Donato S, Zagonel V, Boni L, Falcone A, Danesi R. DPYD and UGT1A1 genotyping to predict adverse events during first-line FOLFIRI or FOLFOXIRI plus bevacizumab in metastatic colorectal cancer. Oncotarget. 2017 Dec 21;9(8):7859-7866. doi: 10.18632/oncotarget.23559. eCollection 2018 Jan 30. PMID 29487697
- [Derived] Cremolini C, Casagrande M, Loupakis F, Aprile G, Bergamo F, Masi G, Moretto R R, Pietrantonio F, Marmorino F, Zucchelli G, Tomasello G, Tonini G, Allegrini G, Granetto C, Ferrari L, Urbani L, Cillo U, Pilati P, Sensi E, Pellegrinelli A, Milione M, Fontanini G, Falcone A. Efficacy of FOLFOXIRI plus bevacizumab in liver-limited metastatic colorectal cancer: A pooled analysis of clinical studies by Gruppo Oncologico del Nord Ovest. Eur J Cancer. 2017 Mar;73:74-84. doi: 10.1016/j.ejca.2016.10.028. Epub 2016 Dec 13. PMID 27986363
- [Derived] Cremolini C, Loupakis F, Masi G, Lonardi S, Granetto C, Mancini ML, Chiara S, Moretto R, Rossini D, Vitello S, Allegrini G, Tonini G, Bergamo F, Tomasello G, Ronzoni M, Buonadonna A, Bustreo S, Barbara C, Boni L, Falcone A. FOLFOXIRI or FOLFOXIRI plus bevacizumab as first-line treatment of metastatic colorectal cancer: a propensity score-adjusted analysis from two randomized clinical trials. Ann Oncol. 2016 May;27(5):843-9. doi: 10.1093/annonc/mdw052. Epub 2016 Feb 9. PMID 26861604
- [Derived] Cremolini C, Loupakis F, Antoniotti C, Lupi C, Sensi E, Lonardi S, Mezi S, Tomasello G, Ronzoni M, Zaniboni A, Tonini G, Carlomagno C, Allegrini G, Chiara S, D'Amico M, Granetto C, Cazzaniga M, Boni L, Fontanini G, Falcone A. FOLFOXIRI plus bevacizumab versus FOLFIRI plus bevacizumab as first-line treatment of patients with metastatic colorectal cancer: updated overall survival and molecular subgroup analyses of the open-label, phase 3 TRIBE study. Lancet Oncol. 2015 Oct;16(13):1306-15. doi: 10.1016/S1470-2045(15)00122-9. Epub 2015 Aug 31. PMID 26338525
- [Derived] Cremolini C, Loupakis F, Antoniotti C, Lonardi S, Masi G, Salvatore L, Cortesi E, Tomasello G, Spadi R, Zaniboni A, Tonini G, Barone C, Vitello S, Longarini R, Bonetti A, D'Amico M, Di Donato S, Granetto C, Boni L, Falcone A. Early tumor shrinkage and depth of response predict long-term outcome in metastatic colorectal cancer patients treated with first-line chemotherapy plus bevacizumab: results from phase III TRIBE trial by the Gruppo Oncologico del Nord Ovest. Ann Oncol. 2015 Jun;26(6):1188-1194. doi: 10.1093/annonc/mdv112. Epub 2015 Feb 23. PMID 25712456
- [Derived] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750